CLINICAL TRIAL: NCT05194722
Title: Optimizing Implementation of Mental Health Intervention Within Orthopedic Care
Brief Title: Optimizing Mental Health in Orthopedic Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Abby Cheng, Assistant Professor, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202110165; P50MH122351 (NIH)
Record Dates: First submitted 2021-12-15; First posted 2022-01-18 (Actual); Results first posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-10

CONDITIONS: Anxiety; Depression; Back Pain; Neck Pain
Keywords: Anxiety; Depression; Spine; Chronic pain; Digital mental health intervention; Orthopedics
MeSH Terms: conditions — Anxiety Disorders; Depression; Back Pain; Neck Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orthopedic spine patients (Experimental): In addition to participating in semi-structured interviews and usability testing of the study interventions, participants in this arm will receive one month of access to Wysa. They will complete measures of clinical effectiveness and hypothesized behavioral targets at baseline and one-month follow-up.
  Interventions: Behavioral: Wysa mobile app

INTERVENTIONS:
Behavioral: Wysa mobile app — Wysa is a digital mental health intervention (i.e., mobile app) that uses an artificial intelligence based chatbot and text-based conversation with master's level human "coach" counselors to deliver cognitive behavioral therapy, mindfulness training, and sleep tools. In this study, a customized version of Wysa will be used which is specifically designed for users with coexisting chronic pain. The customized experience includes additional features based on behavioral activation. This version is not currently commercially available.

SUMMARY:
This study will utilize qualitative cross-sectional and quantitative longitudinal methods. In semi-structured interviews, orthopedic providers and patients with spine conditions will discuss their overall perspectives, specific needs, and preferred solutions to addressing mental health impairment in the context of orthopedic care and research. In these sessions, patient stakeholders will also user test two specific mental health interventions: a customized version of a commercial digital mental health intervention (Wysa) and a prototype of a print-based mental health resource guide. The patient stakeholders will be provided one month of Wysa access, and they will complete baseline and follow-up measures related to usability, clinical effectiveness, and intermediate behavioral mechanisms through which Wysa is hypothesized to act. Wysa usage data will be obtained from the app company. Delivery of Wysa and the printed resource guide will be iteratively refined based on user feedback.

DETAILED DESCRIPTION:
Depression and anxiety heighten musculoskeletal pain and negatively impact outcomes after orthopedic surgery. This phenomenon is especially prevalent in older adults. Our ongoing pilot work demonstrates promise that an established digital mental health intervention (Wysa) can improve orthopedic patients' mental health symptoms, but we also encountered implementation barriers related to discussing mental health in an orthopedic setting. The long-term goal of this line of research is to enable the provision of true comprehensive care to improve both the physical and mental health of orthopedic patients. The goals of this project are to address the implementation barriers we encountered in our ongoing pilot work and to prepare for a definitive trial to assess the effectiveness of a digital mental health intervention in the context of orthopedic care.

The specific aims are to: 1.) identify the contextual determinants of implementation success for addressing patients' mental health in the context of orthopedic care; 2.) conduct usability testing for two mental health interventions which can feasibly be implemented in a real-world orthopedic setting: a digital mental health intervention (Wysa) and a novel printed resource guide; and 3.) identify the intermediate mechanisms through which a digital mental health intervention (Wysa) improves mental health symptoms in orthopedic patients.

Using standard qualitative methods and guided by the Consolidated Framework for Implementation Research (CFIR) and the COM-B model of behavior change, two stakeholder groups will be interviewed: orthopedic providers and older adult orthopedic spine patients. In addition to addressing specific needs and preferences related to discussing mental health in the setting of orthopedic care, patient stakeholders will complete usability testing of Wysa and of the novel printed guide of local and online mental health resources. Next, the patient stakeholders will receive one month of access to Wysa. They will complete measures of clinical effectiveness (self-reported depression, anxiety, pain interference, physical function) and hypothesized behavioral targets (behavioral activation, pain acceptance, sleep quality) at baseline and one-month follow-up. The study findings will facilitate design of a subsequent clinical effectiveness trial that is designed for equitable dissemination and effective implementation of mental health intervention within the context of orthopedic care.

ELIGIBILITY:
Inclusion criteria:

* Orthopedic patient presenting for outpatient clinic evaluation to a spine specialist for neck and/or back pain
* Musculoskeletal spine pain for 3+ months

Exclusion criteria:

* Routine post-operative visit with no plans for further surgery
* Endorses mental health crisis (active suicidal or homicidal ideation, psychosis)
* Cognitive impairment which would interfere with meaningful engagement with research interview, questionnaires, and/or intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-06-18 (Actual); Study Completion 2022-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abby Cheng, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared due to the pilot nature of this study.

REFERENCES:
- [Background] Tunks ER, Crook J, Weir R. Epidemiology of chronic pain with psychological comorbidity: prevalence, risk, course, and prognosis. Can J Psychiatry. 2008 Apr;53(4):224-34. doi: 10.1177/070674370805300403. PMID 18478825
- [Background] Cheng AL, Schwabe M, Doering MM, Colditz GA, Prather H. The Effect of Psychological Impairment on Outcomes in Patients With Prearthritic Hip Disorders: A Systematic Review and Meta-analysis. Am J Sports Med. 2020 Aug;48(10):2563-2571. doi: 10.1177/0363546519883246. Epub 2019 Dec 12. PMID 31829034
- [Background] Edwards RR, Klick B, Buenaver L, Max MB, Haythornthwaite JA, Keller RB, Atlas SJ. Symptoms of distress as prospective predictors of pain-related sciatica treatment outcomes. Pain. 2007 Jul;130(1-2):47-55. doi: 10.1016/j.pain.2006.10.026. Epub 2006 Dec 6. PMID 17156925
- [Background] Lee H, Hubscher M, Moseley GL, Kamper SJ, Traeger AC, Mansell G, McAuley JH. How does pain lead to disability? A systematic review and meta-analysis of mediation studies in people with back and neck pain. Pain. 2015 Jun;156(6):988-997. doi: 10.1097/j.pain.0000000000000146. PMID 25760473
- [Background] Alattas SA, Smith T, Bhatti M, Wilson-Nunn D, Donell S. Greater pre-operative anxiety, pain and poorer function predict a worse outcome of a total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2017 Nov;25(11):3403-3410. doi: 10.1007/s00167-016-4314-8. Epub 2016 Oct 12. PMID 27734110
- [Background] Archer KR, Devin CJ, Vanston SW, Koyama T, Phillips SE, Mathis SL, George SZ, McGirt MJ, Spengler DM, Aaronson OS, Cheng JS, Wegener ST. Cognitive-Behavioral-Based Physical Therapy for Patients With Chronic Pain Undergoing Lumbar Spine Surgery: A Randomized Controlled Trial. J Pain. 2016 Jan;17(1):76-89. doi: 10.1016/j.jpain.2015.09.013. Epub 2015 Oct 23. PMID 26476267
- [Background] la Cour P, Petersen M. Effects of mindfulness meditation on chronic pain: a randomized controlled trial. Pain Med. 2015 Apr;16(4):641-52. doi: 10.1111/pme.12605. Epub 2014 Nov 7. PMID 25376753
- [Background] Kamper SJ, Apeldoorn AT, Chiarotto A, Smeets RJ, Ostelo RW, Guzman J, van Tulder MW. Multidisciplinary biopsychosocial rehabilitation for chronic low back pain: Cochrane systematic review and meta-analysis. BMJ. 2015 Feb 18;350:h444. doi: 10.1136/bmj.h444. PMID 25694111
- [Background] Vranceanu AM, Beks RB, Guitton TG, Janssen SJ, Ring D. How do Orthopaedic Surgeons Address Psychological Aspects of Illness? Arch Bone Jt Surg. 2017 Jan;5(1):2-9. PMID 28271080
- [Background] Andrade LH, Alonso J, Mneimneh Z, Wells JE, Al-Hamzawi A, Borges G, Bromet E, Bruffaerts R, de Girolamo G, de Graaf R, Florescu S, Gureje O, Hinkov HR, Hu C, Huang Y, Hwang I, Jin R, Karam EG, Kovess-Masfety V, Levinson D, Matschinger H, O'Neill S, Posada-Villa J, Sagar R, Sampson NA, Sasu C, Stein DJ, Takeshima T, Viana MC, Xavier M, Kessler RC. Barriers to mental health treatment: results from the WHO World Mental Health surveys. Psychol Med. 2014 Apr;44(6):1303-17. doi: 10.1017/S0033291713001943. Epub 2013 Aug 9. PMID 23931656
- [Background] Kozloff N, Sommers BD. Insurance Coverage and Health Outcomes in Young Adults With Mental Illness Following the Affordable Care Act Dependent Coverage Expansion. J Clin Psychiatry. 2017 Jul;78(7):e821-e827. doi: 10.4088/JCP.16m11357. PMID 28703947
- [Background] Appelbaum PS, Parks J. Holding Insurers Accountable for Parity in Coverage of Mental Health Treatment. Psychiatr Serv. 2020 Feb 1;71(2):202-204. doi: 10.1176/appi.ps.201900513. Epub 2019 Nov 14. PMID 31722647
- [Background] Abraham J, Meng A, Siraco S, Kannampallil T, Politi MC, Baumann AA, Lenze EJ, Avidan MS. A Qualitative Study of Perioperative Depression and Anxiety in Older Adults. Am J Geriatr Psychiatry. 2020 Oct;28(10):1107-1118. doi: 10.1016/j.jagp.2020.02.010. Epub 2020 Mar 2. PMID 32234274
- [Background] Weil TP. Insufficient dollars and qualified personnel to meet United States mental health needs. J Nerv Ment Dis. 2015 Apr;203(4):233-40. doi: 10.1097/NMD.0000000000000271. PMID 25816044
- [Background] Asada Y, Whipp A, Kindig D, Billard B, Rudolph B. Inequalities in multiple health outcomes by education, sex, and race in 93 US counties: why we should measure them all. Int J Equity Health. 2014 Jun 13;13:47. doi: 10.1186/1475-9276-13-47. PMID 24927805
- [Background] Haggerty AF, Hagemann A, Barnett M, Thornquist M, Neuhouser ML, Horowitz N, Colditz GA, Sarwer DB, Ko EM, Allison KC. A Randomized, Controlled, Multicenter Study of Technology-Based Weight Loss Interventions among Endometrial Cancer Survivors. Obesity (Silver Spring). 2017 Nov;25 Suppl 2(Suppl 2):S102-S108. doi: 10.1002/oby.22021. PMID 29086522
- [Background] Cella D, Yount S, Rothrock N, Gershon R, Cook K, Reeve B, Ader D, Fries JF, Bruce B, Rose M; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS): progress of an NIH Roadmap cooperative group during its first two years. Med Care. 2007 May;45(5 Suppl 1):S3-S11. doi: 10.1097/01.mlr.0000258615.42478.55. PMID 17443116
- [Background] Fuhr K, Hautzinger M, Krisch K, Berking M, Ebert DD. Validation of the Behavioral Activation for Depression Scale (BADS)-Psychometric properties of the long and short form. Compr Psychiatry. 2016 Apr;66:209-18. doi: 10.1016/j.comppsych.2016.02.004. Epub 2016 Feb 9. PMID 26995255
- [Background] Fish RA, Hogan MJ, Morrison TG, Stewart I, McGuire BE. Willing and able: a closer look at pain Willingness and Activity Engagement on the Chronic Pain Acceptance Questionnaire (CPAQ-8). J Pain. 2013 Mar;14(3):233-45. doi: 10.1016/j.jpain.2012.11.004. PMID 23452647
- [Background] Fish RA, McGuire B, Hogan M, Morrison TG, Stewart I. Validation of the chronic pain acceptance questionnaire (CPAQ) in an Internet sample and development and preliminary validation of the CPAQ-8. Pain. 2010 Jun;149(3):435-443. doi: 10.1016/j.pain.2009.12.016. Epub 2010 Feb 25. PMID 20188472
- [Background] Baranoff J, Hanrahan SJ, Kapur D, Connor JP. Six month post-treatment deterioration in acceptance (CPAQ-8) and cognitions following multidisciplinary pain treatment. J Behav Med. 2014 Jun;37(3):469-79. doi: 10.1007/s10865-013-9502-0. Epub 2013 Mar 16. PMID 23504128
- [Background] Baranoff J, Hanrahan SJ, Kapur D, Connor JP. Validation of the Chronic Pain Acceptance Questionnaire-8 in an Australian pain clinic sample. Int J Behav Med. 2014 Feb;21(1):177-85. doi: 10.1007/s12529-012-9278-6. PMID 23179676
- [Background] Soldatos CR, Dikeos DG, Paparrigopoulos TJ. The diagnostic validity of the Athens Insomnia Scale. J Psychosom Res. 2003 Sep;55(3):263-7. doi: 10.1016/s0022-3999(02)00604-9. PMID 12932801
- [Background] Soldatos CR, Dikeos DG, Paparrigopoulos TJ. Athens Insomnia Scale: validation of an instrument based on ICD-10 criteria. J Psychosom Res. 2000 Jun;48(6):555-60. doi: 10.1016/s0022-3999(00)00095-7. PMID 11033374
- [Background] Guglielmo D, Hootman JM, Boring MA, Murphy LB, Theis KA, Croft JB, Barbour KE, Katz PP, Helmick CG. Symptoms of Anxiety and Depression Among Adults with Arthritis - United States, 2015-2017. MMWR Morb Mortal Wkly Rep. 2018 Oct 5;67(39):1081-1087. doi: 10.15585/mmwr.mm6739a2. PMID 30286053
- [Background] Murphy LB, Sacks JJ, Brady TJ, Hootman JM, Chapman DP. Anxiety and depression among US adults with arthritis: prevalence and correlates. Arthritis Care Res (Hoboken). 2012 Jul;64(7):968-76. doi: 10.1002/acr.21685. PMID 22550055
- [Background] Bartels SJ, Coakley EH, Zubritsky C, Ware JH, Miles KM, Arean PA, Chen H, Oslin DW, Llorente MD, Costantino G, Quijano L, McIntyre JS, Linkins KW, Oxman TE, Maxwell J, Levkoff SE; PRISM-E Investigators. Improving access to geriatric mental health services: a randomized trial comparing treatment engagement with integrated versus enhanced referral care for depression, anxiety, and at-risk alcohol use. Am J Psychiatry. 2004 Aug;161(8):1455-62. doi: 10.1176/appi.ajp.161.8.1455. PMID 15285973
- [Background] Firth J, Torous J, Nicholas J, Carney R, Rosenbaum S, Sarris J. Can smartphone mental health interventions reduce symptoms of anxiety? A meta-analysis of randomized controlled trials. J Affect Disord. 2017 Aug 15;218:15-22. doi: 10.1016/j.jad.2017.04.046. Epub 2017 Apr 25. PMID 28456072
- [Background] Davies EB, Morriss R, Glazebrook C. Computer-delivered and web-based interventions to improve depression, anxiety, and psychological well-being of university students: a systematic review and meta-analysis. J Med Internet Res. 2014 May 16;16(5):e130. doi: 10.2196/jmir.3142. PMID 24836465
- [Background] Mayberry LS, Lyles CR, Oldenburg B, Osborn CY, Parks M, Peek ME. mHealth Interventions for Disadvantaged and Vulnerable People with Type 2 Diabetes. Curr Diab Rep. 2019 Nov 25;19(12):148. doi: 10.1007/s11892-019-1280-9. PMID 31768662
- [Background] Lee AC, Driban JB, Price LL, Harvey WF, Rodday AM, Wang C. Responsiveness and Minimally Important Differences for 4 Patient-Reported Outcomes Measurement Information System Short Forms: Physical Function, Pain Interference, Depression, and Anxiety in Knee Osteoarthritis. J Pain. 2017 Sep;18(9):1096-1110. doi: 10.1016/j.jpain.2017.05.001. Epub 2017 May 10. PMID 28501708
- [Background] Beleckas CM, Prather H, Guattery J, Wright M, Kelly M, Calfee RP. Anxiety in the orthopedic patient: using PROMIS to assess mental health. Qual Life Res. 2018 Sep;27(9):2275-2282. doi: 10.1007/s11136-018-1867-7. Epub 2018 May 8. PMID 29740783
- [Background] Guattery JM, Dardas AZ, Kelly M, Chamberlain A, McAndrew C, Calfee RP. Floor Effect of PROMIS Depression CAT Associated With Hasty Completion in Orthopaedic Surgery Patients. Clin Orthop Relat Res. 2018 Apr;476(4):696-703. doi: 10.1007/s11999.0000000000000076. PMID 29419628
- [Background] Dy CJ, Brogan DM, Rolf L, Ray WZ, Wolfe SW, James AS. A qualitative study of life satisfaction after surgery for adult traumatic brachial plexus injury. Bone Jt Open. 2021 Jan 3;2(1):9-15. doi: 10.1302/2633-1462.21.BJO-2020-0175.R1. eCollection 2021 Jan. PMID 33537671
- [Background] Dy CJ, Brogan DM, Rolf L, Ray WZ, Wolfe SW, James AS. Variability in Surgeon Approaches to Emotional Recovery and Expectation Setting After Adult Traumatic Brachial Plexus Injury. J Hand Surg Glob Online. 2021 Jan;3(1):30-35. doi: 10.1016/j.jhsg.2020.10.010. Epub 2020 Nov 21. PMID 33537663
- [Background] Prather H, Cheng A, Steger-May K, Maheshwari V, Van Dillen L. Hip and Lumbar Spine Physical Examination Findings in People Presenting With Low Back Pain, With or Without Lower Extremity Pain. J Orthop Sports Phys Ther. 2017 Mar;47(3):163-172. doi: 10.2519/jospt.2017.6567. Epub 2017 Feb 3. PMID 28158964
- [Background] Prather H, Cheng A, Steger-May K, Maheshwari V, VanDillen L. Association of Hip Radiograph Findings With Pain and Function in Patients Presenting With Low Back Pain. PM R. 2018 Jan;10(1):11-18. doi: 10.1016/j.pmrj.2017.06.003. Epub 2017 Jun 16. PMID 28629805
- [Background] Burkhardt HA, Alexopoulos GS, Pullmann MD, Hull TD, Arean PA, Cohen T. Behavioral Activation and Depression Symptomatology: Longitudinal Assessment of Linguistic Indicators in Text-Based Therapy Sessions. J Med Internet Res. 2021 Jul 14;23(7):e28244. doi: 10.2196/28244. PMID 34259637
- [Background] Fortuna KL, Torous J, Depp CA, Jimenez DE, Arean PA, Walker R, Ajilore O, Goldstein CM, Cosco TD, Brooks JM, Vahia IV, Bartels SJ. A Future Research Agenda for Digital Geriatric Mental Healthcare. Am J Geriatr Psychiatry. 2019 Nov;27(11):1277-1285. doi: 10.1016/j.jagp.2019.05.013. Epub 2019 May 23. PMID 31196619
- [Background] Sharpe L, McDonald S, Correia H, Raue PJ, Meade T, Nicholas M, Arean P. Pain severity predicts depressive symptoms over and above individual illnesses and multimorbidity in older adults. BMC Psychiatry. 2017 May 4;17(1):166. doi: 10.1186/s12888-017-1334-y. PMID 28472936
- [Background] Cheng AL, Calfee R, Colditz G, Prather H. PROMIS Physical and Emotional Health Scores Are Worse in Musculoskeletal Patients Presenting to Physiatrists than to Other Orthopedic Specialists. PM R. 2019 Jun;11(6):604-612. doi: 10.1002/pmrj.12068. Epub 2019 Mar 25. PMID 30609319
- [Background] Jensen MP, Ehde DM, Day MA. The Behavioral Activation and Inhibition Systems: Implications for Understanding and Treating Chronic Pain. J Pain. 2016 May;17(5):529.e1-529.e18. doi: 10.1016/j.jpain.2016.02.001. Epub 2016 Mar 24. PMID 27052644
- [Background] Beaton DE, Clark JP. Qualitative research: a review of methods with use of examples from the total knee replacement literature. J Bone Joint Surg Am. 2009 May;91 Suppl 3:107-12. doi: 10.2106/JBJS.H.01631. PMID 19411508
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Derived] Cheng AL, Agarwal M, Armbrecht MA, Abraham J, Calfee RP, Goss CW. Behavioral Mechanisms That Mediate Mental and Physical Health Improvements in People With Chronic Pain Who Receive a Digital Health Intervention: Prospective Cohort Pilot Study. JMIR Form Res. 2023 Nov 17;7:e51422. doi: 10.2196/51422. PMID 37976097

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Orthopedic Spine Patients
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Orthopedic Spine Patients
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (14)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 21
  Sex: Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Adult PROMIS CAT Depression v1.0
Description: The PROMIS (Patient-Reported Outcomes Measurement Information System) Depression measure is a brief, computer-adapted measure of depression symptoms. It is a normalized measure with a mean of 50 and standard deviation of 10. Higher scores represent increased depression symptoms.
Time Frame: Change in score from baseline to post-treatment (Month 1)
Measure: Number (80% Confidence Interval); unit: T-score
Arm/Group | Orthopedic Spine Patients
Number analyzed (Participants) | 30
T-score | -1.3 [-2.9 to 0.3]

2. Primary Outcome: Adult PROMIS CAT Anxiety v1.0
Description: The PROMIS (Patient-Reported Outcomes Measurement Information System) Anxiety measure is a brief, computer-adapted measure of anxiety symptoms. It is a normalized measure with a mean of 50 and standard deviation of 10. Higher scores represent increased anxiety symptoms.
Time Frame: Change in score from baseline to post-treatment (Month 1)
Measure: Mean (80% Confidence Interval); unit: T-score
Arm/Group | Orthopedic Spine Patients
Number analyzed (Participants) | 30
T-score | -3.2 [-4.3 to -2.0]

3. Secondary Outcome: Adult PROMIS CAT Pain Interference v1.1
Description: The PROMIS (Patient-Reported Outcomes Measurement Information System) Pain Interference measure is a brief, computer-adapted measure of how much pain interferes with a person's life. It is a normalized measure with a mean of 50 and standard deviation of 10. Higher scores represent increased pain interference.
Time Frame: Change in score from baseline to post-treatment (Month 1)
Measure: Mean (80% Confidence Interval); unit: T-score
Arm/Group | Orthopedic Spine Patients
Number analyzed (Participants) | 30
T-score | -3.5 [-4.8 to -2.2]

4. Secondary Outcome: Adult PROMIS CAT Physical Function v2.0
Description: The PROMIS (Patient-Reported Outcomes Measurement Information System) Physical Function measure is a brief, computer-adapted measure of a person's self-reported physical functioning. It is a normalized measure with a mean of 50 and standard deviation of 10. Higher scores represent better physical functioning.
Time Frame: Change in score from baseline to post-treatment (Month 1)
Measure: Mean (80% Confidence Interval); unit: T-score
Arm/Group | Orthopedic Spine Patients
Number analyzed (Participants) | 30
T-score | 1.4 [-0.2 to 2.9]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the 1-month intervention time period.
Groups:
- Orthopedic Spine Patients: Orthopaedic spine patients
Arm/Group | Orthopedic Spine Patients
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT05194722/Prot_SAP_000.pdf